CLINICAL TRIAL: NCT02278484
Title: XprESS Device and PathAssist Confirmation Tools in Pediatric Patients-Expanded Indication Study
Brief Title: Sinus Balloon Dilation in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Entellus Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2827-001
Record Dates: First submitted 2014-10-27; First posted 2014-10-30 (Estimated); Results first posted 2016-12-07 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-02

CONDITIONS: Sinusitis
Keywords: sinus infections; sinusitis; chronic sinusitis; rhinosinusitis; allergic sinusitis; allergic rhinitis; chronic rhinosinusitis; sinus disease in children; sinus balloon dilation; balloon dilatation; sinus disease; pediatric
MeSH Terms: conditions — Sinusitis; Rhinosinusitis; Rhinitis, Allergic; Paranasal Sinus Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Balloon Sinus Dilation (Other)
  Interventions: Device: XprESS device and PathAssist confirmation tools

INTERVENTIONS:
Device: XprESS device and PathAssist confirmation tools

SUMMARY:
Safety and effectiveness of sinus balloon dilation in patients 2-21 years old.

ELIGIBILITY:
Inclusion Criteria:

Patients age ≥ 2 to ≤ 21 years old. Diagnosed with Chronic Rhinosinusitis (CRS). Candidate for trans-nasal balloon sinus dilation.

Exclusion Criteria:

History of sinus surgery. Recent nasal or head and neck surgery. Fungal sinus disease. Severe asthma. Cystic fibrosis. Immunodeficiency. Craniofacial abnormalities. Pregnancy (current)

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - North Valley ENT, Phoenix, Arizona
  - Willamette ENT and Facial Plastic Surgery, Salem, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - Alamo ENT and Associates, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Soler ZM, Rosenbloom JS, Skarada D, Gutman M, Hoy MJ, Nguyen SA. Prospective, multicenter evaluation of balloon sinus dilation for treatment of pediatric chronic rhinosinusitis. Int Forum Allergy Rhinol. 2017 Mar;7(3):221-229. doi: 10.1002/alr.21889. Epub 2016 Nov 26. PMID 27888649

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sequential enrollment of eligible participants at sites.
Groups:
- Balloon Sinus Dilation: Balloon Sinus Dilation using XprESS and PathAssist Devices.
Period: Overall Study
Arm/Group | Balloon Sinus Dilation
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Balloon Sinus Dilation
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.7 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 33
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Technical Success: Sinuses Successfully Treated With Balloon Dilation
Description: Number of successful dilations out of all attempted dilations. Success is defined as the device successfully delivered to the target sinus, inflated, deflated, and withdrawn from the treated sinus.
Time Frame: Index procedure
Population: All sinus dilations attempted in all participants
Measure: Number; unit: sinus dilation attempts
Units Other Than Participants: Sinuses
Arm/Group | Balloon Sinus Dilation
Number analyzed (Participants) | 50
Number analyzed (Sinuses) | 157
sinus dilation attempts | 157

2. Primary Outcome: Complications
Description: Number of subjects who experience complications. Complications are defined as serious device or procedure related adverse events.
Time Frame: Index procedure through 3-month follow-up
Population: All participants
Measure: Number; unit: participants
Arm/Group | Balloon Sinus Dilation
Number analyzed (Participants) | 50
participants | 0

3. Secondary Outcome: Change in Quality of Life From Baseline Through Completion
Description: Change in sinonasal symptom severity between the baseline preprocedure assessment and follow-up assessment. Sinus symptom severity is measured using the Sinus and Nasal Quality of Life Survey (SN-5) that is a validated tool for use in pediatric patients (completed by caregivers). The 5 survey items are scored from 1 (best) to 7 (worst) and averaged to provide an overall score.
Time Frame: Baseline to 6-month follow-up
Population: All participants
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Balloon Sinus Dilation
Number analyzed (Participants) | 50
Units on a scale | -2.9 (1.4)
Statistical Analysis 1: Comparison: Balloon Sinus Dilation; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

4. Secondary Outcome: Number of Subjects Who Undergo a Revision or Additional Surgery During the Study
Description: Any surgical intervention that is performed in the sinus(es) following the index procedure will be reported
Time Frame: Procedure-6 month follow up
Population: All participants
Measure: Count of Participants; unit: Participants
Arm/Group | Balloon Sinus Dilation
Number analyzed (Participants) | 50
Participants | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Balloon Sinus Dilation
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less